CLINICAL TRIAL: NCT00551915
Title: Safety, Tolerability, and Immunogenicity of 3 Different Formulations of a Liquid Hexavalent Combination Vaccine, HR5I When Administered to Healthy Hepatitis B Vaccine-Naive Infants at 2, 4, 6, and 12-14 Months of Age
Brief Title: A Study of the Safety and Tolerability of V419 in Healthy Infants at 2,4, 6 and 12 to 14 Months of Age (V419-003)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V419-003; 2007_581 (Other: Merck Registration Number)
Record Dates: First submitted 2007-10-29; First posted 2007-10-31 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Bacterial Infections; Virus Diseases
MeSH Terms: conditions — Bacterial Infections; Virus Diseases | interventions — pentacel; Recombivax HB

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AR51 (12, 10) (Experimental): Participants were vaccinated with 0.5 ml of AR51 (12,10) formulation via intramuscular injection as a primary series at 2, 4, and 6 months of age, and as a booster at 12 to 14 months of age.
  Interventions: Biological: AR51 (12, 10)
- PR51 (3, 10) (Experimental): Participants were vaccinated with 0.5 ml of PR51 (3,10) formulation via intramuscular injection as a primary series at 2, 4, and 6 months of age, and as a booster at 12 to 14 months of age.
  Interventions: Biological: PR51 (3, 10)
- PR51 (6, 10) (Experimental): Participants were vaccinated with 0.5 ml of PR51 (6,10) formulation via intramuscular injection as a primary series at 2, 4, and 6 months of age, and as a booster at 12 to 14 months of age.
  Interventions: Biological: PR51 (6, 10)
- PENTACEL™ + RECOMBIVAX HB™ (Active Comparator): Participants were vaccinated with 0.5 ml each of PENTACEL™ + RECOMBIVAX HB™ via intramuscular injection as a primary series at 2, 4, and 6 months of age, and with 0.5 ml PENTACEL™ as a booster at 12 to 14 months of age.
  Interventions: Biological: PENTACEL™; Biological: RECOMBIVAX HB™

INTERVENTIONS:
Biological: AR51 (12, 10) — vaccine formulation containing 12 mcg of PRP-T and 10 mcg of HBsAg
  Arms: AR51 (12, 10)
Biological: PR51 (3, 10) — vaccine formulation containing 3 mcg of PRP-OMPC and 10 mcg of HBsAg
  Arms: PR51 (3, 10)
Biological: PR51 (6, 10) — vaccine formulation containing 6 mcg of PRP-OMPC and 10 mcg of HBsAg
  Arms: PR51 (6, 10)
Biological: PENTACEL™ — licensed vaccine for diphtheria, tetanus, pertussis, poliomyelitis, and invasive disease due to Haemophilus influenzae type b, administered open-label
  Arms: PENTACEL™ + RECOMBIVAX HB™
Biological: RECOMBIVAX HB™ — licensed vaccine for hepatitis, administered open-label
  Arms: PENTACEL™ + RECOMBIVAX HB™

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and immunogenicity of 3 formulations of the HR5I vaccine (Haemophilus influenzae type b conjugate, recombinant hepatitis B surface antigen, diphtheria, tetanus, 5-component acellular pertussis, and inactivated poliovirus Types 1, 2, and 3). The primary hypothesis is that at least 1 of the 3 formulations of HR5I administered as a primary series at 2, 4, and 6 months of age will be acceptable (similar to targeted rates) with respect to Postdose 3 antibody responses to all antigens.

DETAILED DESCRIPTION:
Participants will be randomized into 4 arms:

AR51 (12, 10): arm receiving vaccine formulation containing 12 mcg of polyribosylribitol phosphate (PRP) conjugated to tetanus toxoid (PRP-T) and 10 mcg of Hepatitis B surface antigen (HBsAg)

PR51 (3, 10): arm receiving vaccine formulation containing 3 mcg of polyribosylribitol phosphate conjugated to the outer membrane protein complex of Neisseria meningitides (PRP-OMPC) and 10 mcg of HBsAg

PR51 (6, 10): arm receiving vaccine formulation containing 6 mcg of PRP-OMPC and 10 mcg of HBsAg

PENTACEL™ + RECOMBIVAX HB™: open-label control group receiving PENTACEL™ (licensed vaccine for diphtheria, tetanus, pertussis, poliomyelitis, and invasive disease due to Haemophilus influenzae type b) and RECOMBIVAX HB™ (licensed vaccine for hepatitis)

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants 2 months of age who have not received prior vaccinations for Haemophilus influenzae type b (Hib), hepatitis B, Diptheria/Pertussis/Tetanus (DPT), or Polio

Exclusion Criteria:

* HIV infection in participant (child/mother)
* Documented HBsAg seropositivity in the participant (child or mother)
* History of invasive Hib disease, hepatitis B, diphtheria, tetanus, pertussis, or poliovirus infection
* History of seizure disorder
* Underlying medical conditions such as inborn errors of metabolism, failure to thrive, or any major congenital abnormalities requiring surgery
* Prior or anticipated receipt of immune globulin, blood, or blood products
* Known hypersensitivity to any component of the investigational or marketed vaccines being administered in this protocol
* Any history or condition that would exclude the participant from receiving any vaccine administered under this protocol based on the contraindications that appear in the package circulars for each component of these vaccines
* Any condition that, in the opinion of the investigator, is not stable or may interfere with the evaluation of the study objectives

Ages: 6 Weeks to 9 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 756 (Actual)
Dates: Start 2001-05; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with level of anti-PRP antibodies >1.0 μg/mL at the Postdose 3 time point | At 7 months of age (1 month after 3rd vaccination)
Percentage of participants with level of anti-HBsAg antibodies ≥10 mIU/L at the Postdose 3 time point | At 7 months of age (1 month after 3rd vaccination)
Percentage of participants with a ≥4-fold rise in levels of antibodies to pertussis antigens at the Postdose 3 time point | At 7 months of age (1 month after 3rd vaccination)
Percentage of participants with level of anti-diphtheria antibodies ≥0.01 IU/mL at the Postdose 3 time point | At 7 months of age (1 month after 3rd vaccination)
Percentage of participants with level of anti-tetanus antibodies ≥0.01 IU/mL at the Postdose 3 time point | At 7 months of age (1 month after 3rd vaccination)
Percentage of participants with neutralizing anti-poliovirus type antibodies at ≥1:8 dilution at the Postdose 3 time point | At 7 months of age (1 month after 3rd vaccination)

SECONDARY OUTCOMES:
Percentage of participants with level of anti-PRP antibodies >1.0 μg/mL at the Postdose 2 time point | At 6 months of age (2 months after 2nd vaccination)
Percentage of participants with level of anti-HBsAg antibodies ≥10 mIU/L at the Postdose 2 time point | At 6 months of age (2 months after 2nd vaccination)
Percentage of participants with a ≥4-fold rise in level of antibodies to pertussis antigens at the Postdose 2 time point | At 6 months of age (2 months after 2nd vaccination)
Percentage of participants with level of anti-diphtheria antibodies ≥0.01 IU/mL at the Postdose 2 time point | At 6 months of age (2 months after 2nd vaccination)
Percentage of participants with level of anti-tetanus antibodies ≥0.01 IU/mL at the Postdose 2 time point | At 6 months of age (2 months after 2nd vaccination)
Percentage of participants with neutralizing anti-poliovirus type antibodies at ≥1:8 dilution at the Postdose 2 time point | At 6 months of age (2 months after 2nd vaccination)
Number of participants with at least 1 adverse event (AE) | From 1st vaccination up to 14 days following last vaccination (up to 14.5 months)
Number of participants who discontinued study treatment due to an AE | From 1st vaccination up to 14 days following last vaccination (up to 14.5 months)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Diaz-Mitoma F, Halperin SA, Tapiero B, Hoffenbach A, Zappacosta PS, Radley D, Bradshaw S, Martin JC, Boslego JW, Hesley TM, Bhuyan PK, Silber JL. Safety and immunogenicity of three different formulations of a liquid hexavalent diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine at 2, 4, 6 and 12-14 months of age. Vaccine. 2011 Feb 1;29(6):1324-31. doi: 10.1016/j.vaccine.2010.11.053. Epub 2010 Dec 4. PMID 21134456